CLINICAL TRIAL: NCT02515422
Title: Subcutaneous Wound Infiltration of Ketamine is Superior to Bupivacaine in Terms of Pain Perception and Opioid Consumption After Cesarean Section: a Double-blinded Randomized Placebo Controlled Clinical Trial.
Brief Title: Subcutaneous Wound Infiltration of Ketamine or Bupivacaine Pain Perception After Cesarean Section
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huseyin Aksoy (Other Government)
Responsible Party: Sponsor-Investigator, Huseyin Aksoy, M.D., Kayseri Education and Research Hospital
Organization: Kayseri Education and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2014/99
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Postoperative Pain
Keywords: Caesarean Section
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Group 1, Ketamine (Active Comparator): Ketamine, 1 mg/kg (Ketalar®, 10 mL inj., 50 mg ketamine hydrochloride/ml, Pfizer Drug Company, USA) was administered subcutaneously before the closure of pfannenstiel incision.
  Interventions: Drug: Ketamine
- Group 2, Bupivacaine (Active Comparator): Bupivacaine 0.5% 20 mL (100 mg) (Marcaine®, 20 mL inj. 5 mg bupivacaine hydrochloride/ml, AstraZeneca Drug Company, Turkey) was administered subcutaneously before the closure of pfannenstiel incision.
  Interventions: Drug: Bupivacaine
- Group 3, Ketamine+Bupivacaine (Active Comparator): Ketamine 1 mg/kg (Ketalar®) and bupivacaine 0.5% (100 mg) (Marcaine®) were administered subcutaneously before the closure of pfannenstiel incision.
  Interventions: Drug: Ketamine; Drug: Bupivacaine
- Group 4, Placebo (Placebo Comparator): Placebo (0.9% saline solution) was administered subcutaneously before the closure of pfannenstiel incision.
  Interventions: Drug: Placebo (0.9% saline solution)

INTERVENTIONS:
Drug: Ketamine — Subcutaneous infiltration of ketamine
  Other Names: Ketalar
  Arms: Group 1, Ketamine; Group 3, Ketamine+Bupivacaine
Drug: Bupivacaine — Subcutaneous infiltration of bupivacaine
  Other Names: Marcaine
  Arms: Group 2, Bupivacaine; Group 3, Ketamine+Bupivacaine
Drug: Placebo (0.9% saline solution)
  Arms: Group 4, Placebo

SUMMARY:
Aim: To assess the analgesic efficacy of subcutaneous infiltration of ketamine, either alone or as an adjuvant to bupivacaine, following CS and to compare their effects on postoperative pain scores and opioid consumption.

Methods: Included patients were allocated to four treatment groups using computer-generated randomization number chart as follows; Group 1 (Ketamine, n=30) received subcutaneous infiltration of ketamine, Group 2 (Bupivacaine, n=30) received subcutaneous infiltration of bupivacaine 0.5%, Group 3 (Ketamine+Bupivacaine, n=30) received subcutaneous infiltration of ketamine+bupivacaine 0.5% and Group 4 (Placebo, n=30) received subcutaneous infiltration of placebo (0.9% saline solution). Patients, anesthetist, surgeon, and other medical and nursing staff were blinded to the contents of the medications. VAS scores at resting and on coughing and analgesic consumptions were compared.

DETAILED DESCRIPTION:
the Group 1 (Ketamine, n=30) received subcutaneous infiltration of ketamine 1 mg/kg (Ketalar®, 10 mL inj., 50 mg ketamine hydrochloride/ml, Pfizer Drug Company, USA). The Group 2 (Bupivacaine, n=30) received subcutaneous infiltration of 20 mL (100 mg) of bupivacaine 0.5% (Marcaine®, 20 mL inj. 5 mg bupivacaine hydrochloride/ml, AstraZeneca Drug Company, Turkey). The Group 3 (Ketamine+Bupivacaine, n=30) received subcutaneous infiltration of ketamine 1 mg/kg (Ketalar®) plus subcutaneous infiltration of 20 mL (100 mg) of bupivacaine 0.5% (Marcaine®). The Group 4 (Placebo, n=30) received subcutaneous infiltration of 30 mL placebo (0.9% saline solution). All medications were diluted with sterile 0.9% saline solution to 30 ml solutions in the similar volume and shape syringes and were infiltrated subcutaneously along the skin wound edges and close to the fascia prior to skin closure. There were four separate syringes which were prepared by an anesthesiology technician for four different treatment groups labeled G1, G2, G3 and G4 containing the ketamine, bupivacaine, ketamine plus bupivacaine and normal saline solution. Patients, anesthetist, surgeon, and other medical and nursing staff were blinded to the contents of the medications.

ELIGIBILITY:
Inclusion Criteria:

* singleton term pregnancy,
* between 38-41th weeks of gestation,
* absence of any medical or obstetrical problems.

Exclusion Criteria:

* multiple pregnancies,
* intrauterine fetal deaths,
* active stage of labor,
* obstetric emergencies such as antepartum hemorrhage, eclampsia and acute fetal distress,
* special request for general anesthesia,
* history of allergic reaction or sensitivity to any of the drugs used in the study,
* reflected anxiety and depression during the cesarean operation,
* any systemic diseases (chronic hypertension, thyroid diseases, renal or hepatic insufficiency, psychiatric disorders,
* chronic pain syndrome, epilepsy or intracranial hypertension)
* medications that would affect the perception of pain,
* current or past history of narcotic use or a history of narcotic abuse,
* inability to understand how to score a 10-cm visual analogue scale (VAS) for pain.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Postoperative visual analog scale pain score | Postoperative 12 hours

SECONDARY OUTCOMES:
Postoperative opioid consumption | Postoperative 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Educational and Research Hospital, Kayseri, Turkey (Türkiye)